CLINICAL TRIAL: NCT05182281
Title: The Effect of Horizontal Whole-body Vibration Therapy on Bone, Quality of Life, Pain, and Balance in Post-menopausal Women
Brief Title: The Effect of Horizontal Whole-body Vibration Therapy in Post-menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: feyzaakan
Record Dates: First submitted 2021-12-17; First posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Osteoporosis; Whole Body Vibration
Keywords: Osteoporosis; Whole-body vibration; Bone mineral density; Quality of life
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whole Body Vibration and Infrared Therapy Group (Experimental): Patients in the whole body vibration and infrared group received vibration therapy with a frequency of 60 Hz and amplitude of 0.5-2 mm and infrared therapy at a wavelength of 550-950 nm 20 minutes daily session, 2 days per weeks for 3 months.1000 mg Ca and 880 IU vitamin D treatment were given.
  Interventions: Device: Whole Body Vibration and Infrared Therapy
- Infrared Therapy Group (Active Comparator): Patients in infrared therapy group received infrared therapy at a wavelength of 550-950 nm 20 minutes daily session, 2 days per weeks for 3 months.1000 mg Ca and 880 IU vitamin D treatment were given.
  Interventions: Device: Infrared Therapy
- Classical Treatment Group (Other): 1000 mg Ca and 880 IU vitamin D treatment were given.
  Interventions: Other: Classical Treatment

INTERVENTIONS:
Device: Whole Body Vibration and Infrared Therapy — Patients in the whole body vibration and infrared group received vibration therapy with a frequency of 60 Hz and amplitude of 0.5-2 mm and infrared therapy at a wavelength of 550-950 nm. Whole body vibration and infrared treatment were applied with the Power Andullator (HHP, CE0197, Germany) device.
  Arms: Whole Body Vibration and Infrared Therapy Group
Device: Infrared Therapy — Patients in infrared therapy group received infrared therapy at a wavelength of 550-950 nm.Infrared treatment were applied with the Power Andullator (HHP, CE0197, Germany) device.
  Arms: Infrared Therapy Group
Other: Classical Treatment — 1000 mg Ca and 880 IU vitamin D treatment were given
  Arms: Classical Treatment Group

SUMMARY:
Osteoporosis is an important public health issue that may result in a high fracture risk in the elderly population. There is general consensus that physical exercise decreases the risk of osteoporotic fractures by reducing the risk of falls and increasing bone strength. Although long-term high-intensity exercise programs have been shown to be successful in early post-menopausal women, a high-intensity exercise program appears to be less attractive to older post-menopausal women and may cause a lack of compliance in the long term and result in injury. Some studies have described falls and fractures as side effects of exercise.Whole-body vibration (WBV) therapy is an easy-to-apply alternative therapy for those who do not wish to initiate or continue pharmacological treatments and cannot perform high-impact exercises and is associated with high patient compliance. WBV therapy is among the promising new interventions for the prevention and treatment of osteoporosis and is defined as mechanical vibration applied in a standing or supine position without any restrictions on frequency (hertz), amplitude (millimeters), magnitude (vibration acceleration due to gravity, g) and cumulative WBV dose. The evidence obtained from animal studies have shown that WBV can be an effective method for increasing bone mass and improving bone structure and strength. Some human studies have shown that WBV can positively affect BMD and improve neuromuscular parameters associated with falls in post-menopausal women.Small changes in posture can have a significant effect on the extent to which a plantar-based mechanical stimulus is actually transmitted to the spine or hip; the stimulus is likely to be weakened by the inevitable changes in posture, which occur due to aging and osteoporosis. For these reasons, we aimed to examine the effect of high frequency and low-magnitude horizontal vibration therapy in post-menopausal women without being affected by posture in the present study.

DETAILED DESCRIPTION:
In this prospective, randomized controlled 3-month study, 185 post-menopausal women who were diagnosed with osteoporosis and followed up in our outpatient clinic based on the osteoporosis diagnostic criteria by the World Health Organization were analyzed.According to the inclusion and exclusion criteria, 60 patients were included in the study.

The patients included in the study were randomized by the co-researcher into 3 groups of 20 patients each according to the random numbers table. Group 1 received WBV and infrared therapy for 20 minutes per session, 2 days a week for 3 months. Group 2 received only infrared therapy for 20 minutes, 2 days a week for 3 months, in the same bed system. The patients were placed in the supine position with the whole body in contact with the platform/bed during the treatment. In terms of compliance with the WBV therapy, the frequency was increased to 30 Hz in the first week, 40 Hz in the second week, 50 Hz in the third week, and 60 Hz in the fourth week and administered for a total of 20 minutes. Subsequent sessions continued with 60 Hz. The acceleration value administered by the device was 2.0-4.0 m/s², and the amplitude of the applied vibration in the vertical direction was 0.5-2.0 mm.Infrared therapy at a wavelength of 550-950 nm was applied to both groups of patients by means of infrared pads on the bed during the treatment.Group 3 did not receive any treatment. Patients in all 3 groups continued their treatment with 1000 mg Ca and 880 IU vitamin D. The patients were called every week by phone to check whether they were complying with the treatment or not.Bone mineral density (BMD) of the lumbar and femoral regions of all the patients was measured using dual energy x-ray absorptiometry. In addition, osteocalcin and hydroxyproline values were measured. Quality of life was assessed using the Short Form-36 questionnaire, pain was assessed using the visual analog scale, and balance was assessed based on the participants' performance in the Berg Balance test.The scales were applied at the beginning and at the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal female patients
* Aged 45-65 years
* L2-L4 and/or femoral neck BMD T-scores of -2.5 to-3.

Exclusion Criteria:

* Osteoporotic fractures
* Metabolic bone disease
* Hyperparathyroidism
* Presence of hyperthyroidism
* History of steroids or current use of steroids
* History of bisphosphonate consumption over the previous year
* Women with lumbar disk herniation, spondylolisthesis or narrow spinal canal
* Conditions that constitute a contraindication for vibration therapy;
* Kidney stones
* Gallstones
* Pregnancy
* Epilepsy
* Cancer
* Pacemaker
* Treatment of orthostatic hypotension
* Recent implants (joint, cochlear, or corneal)
* Recent surgery
* Recent intrauterine device
* Acute thrombosis or hernia
* Acute rheumatoid arthritis
* Serious cardiovascular event
* Diabetes
* Migraine

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2015-08-01 (Actual); Study Completion 2015-08-01 (Actual)

PRIMARY OUTCOMES:
Body Mass Density | 3 months
  BMD (g/cm²) of the lumbar, femoral neck, and entire femoral regions of all patients was measured at the onset and end of the treatment using dual energy x-ray absorptiometry (General Electric LUNAR Prodigy Advance).
Bone Turnover Markers | 3 months
  Serum samples were taken from all patients between 08:00 and 10:00 in the morning after 12 hours of fasting. Urine samples were analyzed in the first morning urine. We checked the values of osteocalcin (OC) as a bone formation marker and hydroxyproline/creatinine values as a bone resorption marker.
The Short Form-36 | 3 months
  The Short Form-36 (SF-36) is a widely used health-related quality of life scale. It is not specific to any age, disease, or treatment group. It includes general health concepts. It is a questionnaire containing 36 questions in 8 subscales. SF-36 scale can be examined under 2 main sections as physical and mental health. Patients are scored out of 100 points in the SF-36 scale and the scores obtained vary between 0 and 100 points for each component. High scores on this scale indicate a better level of health, whereas low scores indicate deterioration of health.
Visual analog scale | 3 months
  Pain was evaluated according to the visual analog scale (0: no pain; 10 very severe pain). They were asked to describe their back pain on the scale choosing a number from 0 to 10 (10-cm VAS).
Berg Balance Test | 3 months
  Berg Balance test (BBT) assesses whether people can maintain their balance during 14 different activities. The level of competence in the activity for each item is scored between 0 and 4 with 0 indicating the lowest score (incapable of doing) and 4 indicating the highest score (doing it independently and safely). The maximum score obtainable is 56. Higher scores indicate better balance .

CONTACTS AND LOCATIONS:
Overall Officials: Feyza Akan Begoğlu, Principal Investigator — Fatih Sultan Mehmet Training and Research Hospital
Locations (1):
- Feyza Akan BEGOGLU, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No